CLINICAL TRIAL: NCT02241486
Title: A Randomized, Double-blind, Placebo-controlled, Cross-over Trial of Sublingual Fentanyl Spray (Subsys) and Oral Morphine for Procedural Wound Care in Adult Patients With Burn Injury Pain
Brief Title: Sublingual Fentanyl and Procedural Burn Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: No funding source.
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Joseph Holtman, Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 205025
Record Dates: First submitted 2013-11-12; First posted 2014-09-16 (Estimated); Results first posted 2017-06-09 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-06

CONDITIONS: Burn Pain
Keywords: Burn pain; Procedural pain; Sublingual fentanyl; Morphine
MeSH Terms: conditions — Pain; Pain, Procedural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sublingual Fentanyl Spray (Experimental): Examine the efficacy and safety of sublingual fentanyl spray (Subsys) for procedural pain (dressing changes/minor debridement) in patients with burn injury.
  Interventions: Drug: Sublingual Fentanyl Spray

INTERVENTIONS:
Drug: Sublingual Fentanyl Spray — Patients with burn injuries will receive sublingual fentanyl spray (Subsys) for procedural pain (dressing changes/minor debridement).

SUMMARY:
The purpose of this study is to examine the efficacy and safety of sublingual fentanyl spray (Subsys) for procedural pain (dressing changes/minor debridement) in patients with burn injury.

DETAILED DESCRIPTION:
The purpose of this study is to examine the efficacy and safety of sublingual fentanyl spray (Subsys) for procedural pain (dressing changes/minor debridement) in patients with burn injury. It will be compared with a standard treatment regimen of oral morphine. The hypothesis is that the fentanyl spray will be more effective for the treatment of procedural pain in patients with burn injury.

ELIGIBILITY:
Inclusion Criteria:

* Subject capable of giving consent
* Age 18-65
* Total burn surface area greater than or equal to 5%
* Opioid tolerant
* BMI less than or equal to 35

Exclusion Criteria:

* Subjects with cognitive or psychiatric impairment that would preclude study participation or compliance with protocol
* Allergy to fentanyl, morphine, naloxone
* Pregnancy, intent to become pregnant or lactating
* Evidence of burn injury to oral mucosa
* Active illicit drug use or illicit drug abuse history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph R Holtman Jr, MD Ph.D., Principal Investigator — Department Anesthesiology Loyola University Medical Center
Locations (1):
- Loyola University Medical Center Burn Unit, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There are no pre-assignment details.
Period: Overall Study
Arm/Group | Sublingual Fentanyl Spray
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Only two patients were initially enrolled in this trial, which was terminated prematurely.
Arm/Group | Sublingual Fentanyl Spray
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain Relief
Description: Patients suffering from burn injuries will receive sublingual fentanyl spray (Subsys) to address procedural pain (dressing changes/minor debridement). It will be compared with a standard treatment regimen of oral morphine. The hypothesis is that the fentanyl spray will be more effective for the treatment of procedural pain in patients with burn injury.
Time Frame: 60 min
Population: No participants are included in this analysis because the trial was terminated prematurely. As a result, data to assess primary and secondary study aims are incomplete or entirely unavailable for summary or statistical comparisons.
Arm/Group | Sublingual Fentanyl Spray
Number analyzed (Participants) | 0
Value | 0

ADVERSE EVENTS:
Arm/Group | Sublingual Fentanyl Spray
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
This trial was terminated prematurely due to a lack of study funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes